CLINICAL TRIAL: NCT04136925
Title: Evaluation of the Preparation of Runners and the Impact of an Ultra-trail Event in a Hot and Humid Environment (Ultra Trail Adaptation Environment)
Brief Title: Evaluation of the Preparation of Runners and the Impact of an Ultra-trail Event in a Hot and Humid Environment
Acronym: ERUPTION1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/CHU/08
Record Dates: First submitted 2019-10-11; First posted 2019-10-23 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-10

CONDITIONS: Intensive Sport
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- runner participating of the "Grand Raid"
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire before and after race

SUMMARY:
Human beings are characterized by their extraordinary ability to thermoregulate. During a physical exercise, only 25% of the energy provided by the substrates is converted into muscular mechanical work. The remaining 75% is released as heat.

In fact, thermoregulation has always been an integral part of exercise's physiology.

Due to current climate change, study and understand the mechanisms of thermoregulation and the practices of runners to cope with these constraints becomes increasingly necessary in order to optimize the sports performance and protect the health of athletes of all levels.

Heat stroke is responsible for more deaths than any other environmental disaster and is the second leading cause of sport mortality after heart problems.

The exercise-related hyperthermia and malignant hyperthermia, dehydration and hyponatremia problems have been relatively well studied in several sports. For ultra endurance disciplines, the data remains very fragmentary.

ELIGIBILITY:
Inclusion Criteria:

* All major runners participating in one of the 3 individual races of the "Grand Raid" 2019 in Reunion Island

Exclusion Criteria:

* Refusal to participate
* Runners who do not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Runners participating in one of the 3 individual races of the "Grand Raid" 2019 in Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Repercussion of the race on health evaluate by proportion of heat symptoms on our sample | during the 3 days of the race

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOUSCAREN, Principal Investigator — Centre Hospitalier Universitaire de La REUNION
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: Undecided